CLINICAL TRIAL: NCT00513799
Title: The Natural History of Community-Associated Methicillin-Resistant Staphylococcus Aureus (CA-MRSA) Infections and an Evaluation of Decolonization Strategies
Brief Title: The Natural History of Community-Associated MRSA Infections and Decolonization Strategies
Acronym: StLStaRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Stephanie A. Fritz, Assistant Professor of Pediatrics, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9000C4
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Results first posted 2011-03-29 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Abscesses; Furunculosis; Staphylococcus Aureus; Staphylococcal Skin Infections
MeSH Terms: conditions — Abscess; Furunculosis; Staphylococcal Infections; Staphylococcal Skin Infections | interventions — Mupirocin; chlorhexidine gluconate; Indicator Dilution Techniques; Sodium Hypochlorite

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1: Hygiene Education (Active Comparator): Intensive education on prevention of skin infections through improvements in personal hygiene (also serves as "control group")
  Interventions: Behavioral: Intensive education on personal hygiene
- 2: Hygiene education + mupirocin (Active Comparator): Application of mupirocin in the nasal mucosa alone
  Interventions: Drug: Mupirocin ointment; Behavioral: Intensive education on personal hygiene
- Education + mupirocin + chlorhexidine (Active Comparator): A combination of nasal application of mupirocin and chlorhexidine showers
  Interventions: Drug: Mupirocin ointment; Genetic: Chlorhexidine showers; Behavioral: Intensive education on personal hygiene
- 4: Education + mupirocin + bleach baths (Active Comparator): A combination of nasal application of mupirocin and bathing in dilute bleach water
  Interventions: Drug: Mupirocin ointment; Procedure: Bleach baths (dilute); Behavioral: Intensive education on personal hygiene

INTERVENTIONS:
Drug: Mupirocin ointment — Add a small amount of Mupirocin to the cotton end of a swab. Swab in inner nostril, then repeat in other nostril using new cotton swab with ointment. Twice daily treatment for 5 days.
  Other Names: Bactroban
  Arms: 2: Hygiene education + mupirocin; 4: Education + mupirocin + bleach baths; Education + mupirocin + chlorhexidine
Genetic: Chlorhexidine showers — Apply Clorhexidine wash to entire body once daily for 5 days.
  Other Names: Hibiclens
  Arms: Education + mupirocin + chlorhexidine
Procedure: Bleach baths (dilute) — Pour 2 ounces of bleach into water-filled bath tub. Soak in bath for 15 minutes. Apply once daily for 5 days.
  Other Names: Clorox
  Arms: 4: Education + mupirocin + bleach baths
Behavioral: Intensive education on personal hygiene — Repeat hygiene methods for 5 days.

SUMMARY:
The purpose of this study is to determine the natural history of community-associated Staphylococcus aureus infections in both adult and pediatric patients by monitoring the rate of recurrent infections in those colonized with S. aureus.

In addition, this study will evaluate the efficiency of commonly prescribed decolonization measures in patients presenting with S. aureus skin and soft tissue infections.

DETAILED DESCRIPTION:
Infections with community-associated methicillin-resistant Staphylococcus aureus (CA-MRSA) range in severity from superficial skin abscesses to invasive soft tissue infections like cellulitis and pyomyositis. There has been a large increase in the number of patients presenting to our institution with CA-MRSA infections. Colonization with S. aureus (SA) may be linked to the development of infection but data on this phenomenon are limited. The recurrence rate for CA-MRSA soft tissue infections is unknown. A variety of decolonization strategies have been used for infection prophylaxis with varying results, primarily in patients undergoing hemodialysis or surgery. This study seeks to determine the recurrence rate of soft tissue infections among patients with CA-MRSA infections and to determine a reasonable and efficacious decolonization strategy to eradicate CA-MRSA from previously infected patients.

The proposed methods for decolonization will be tested in a randomized controlled trial with four intervention arms. The intervention arms are: (1) intensive education on prevention of skin infections through improvements in personal hygiene (also serves as "control group"), (2) application of mupirocin in the nasal mucosa alone, (3) a combination of nasal application of mupirocin and chlorhexidine showers, and (4) a combination of nasal application of mupirocin and bathing in dilute bleach water. The "control" group as well as the three other arms will receive intensive hygiene education.

Decolonization with mupirocin ointment and chlorhexidine showers or dilute bleach baths in combination are likely to be more successful than either the application of nasal mupirocin ointment alone or hygiene measures alone. It is expected that these decolonization methods will result in a 50% relative reduction in MRSA colonization at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who presents with at least one serious skin or soft tissue infection requiring incision and drainage at an affiliated institution or clinic in the St. Louis metropolitan area

Exclusion Criteria:

* Patients with permanent indwelling catheters or percutaneous medical devices
* Patients with a history of dialysis treatments, long term care facility admission, or presents with a surgical wound infection within the past year
* Patients who are pregnant

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2007-03; Primary Completion 2009-06 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard C. Camins, MD, MSCR, Principal Investigator — Assistant Professor of Medicine, Division of Infectious Diseases, Department of Medicine, Washington University School of Medicine; Gregory A. Storch, MD, Principal Investigator — Professor of Medicine and Molecular Microbiology, Chief of Division of Pediatric Infectious Diseases, Department of Medicine, Washington University School of Medicine
Locations (2):
- United States (2):
  - Barnes-Jewish Hospital, St Louis, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri

REFERENCES:
- [Derived] Fritz SA, Camins BC, Eisenstein KA, Fritz JM, Epplin EK, Burnham CA, Dukes J, Storch GA. Effectiveness of measures to eradicate Staphylococcus aureus carriage in patients with community-associated skin and soft-tissue infections: a randomized trial. Infect Control Hosp Epidemiol. 2011 Sep;32(9):872-80. doi: 10.1086/661285. PMID 21828967

RESULTS

PARTICIPANT FLOW:
Groups:
- Hygiene Education: Participants only administered an intensive education on prevention of skin infections through improvements in personal hygiene (also serves as "control group")
- Hygiene Education + Mupirocin: Participants administered an intensive education on prevention of skin infections through improvements in personal hygiene AND prescribed Mupirocin ointment applied to the nasal mucosa twice daily for 5 days
- Education + Mupirocin + Chlorhexidine: Participants administered an intensive education on prevention of skin infections through improvements in personal hygiene AND prescribed Mupirocin ointment applied to the nasal mucosa twice daily for 5 days AND prescribed Chlorhexidine wash to entire body once daily for 5 days.
- Education + Mupirocin + Bleach Baths: Participants administered an intensive education on prevention of skin infections through improvements in personal hygiene AND prescribed Mupirocin ointment applied to the nasal mucosa twice daily for 5 days AND prescribed bleach bath to entire body once daily for 5 days (instructed to pour 2 ounces of bleach into water-filled bath tub and soak in bath for 15 minutes).
Period: One-Month Follow-Up
Arm/Group | Hygiene Education | Hygiene Education + Mupirocin | Education + Mupirocin + Chlorhexidine | Education + Mupirocin + Bleach Baths
Started | 75 | 75 | 75 | 75
Completed | 64 | 62 | 64 | 54
Not Completed | 11 | 13 | 11 | 21
Period: Four-Month Follow-Up
Arm/Group | Hygiene Education | Hygiene Education + Mupirocin | Education + Mupirocin + Chlorhexidine | Education + Mupirocin + Bleach Baths
Started | 64 | 62 | 64 | 54
Completed | 64 | 57 | 57 | 51
Not Completed | 0 | 5 | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hygiene Education | Hygiene Education + Mupirocin | Education + Mupirocin + Chlorhexidine | Education + Mupirocin + Bleach Baths | Total
Number analyzed (Participants) | 75 | 75 | 75 | 75 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.37 (16.57) | 16.52 (16.12) | 18.19 (17.37) | 18.67 (15.29) | 17.61 (16.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 37 | 52 | 38 | 161
  Male | 41 | 38 | 23 | 37 | 139

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Eradicated of S. Aureus Carriage - 1 Month After Intervention
Description: Eradication is defined as the absence of S. aureus carriage at the 3 sampled body sites (anterior nares, axilla, inguinal folds) of the index patient. Samples obtained by study team at follow-up visit.
Time Frame: 1 month follow-up
Measure: Number; unit: Participants
Arm/Group | Hygiene Education | Hygiene Education + Mupirocin | Education + Mupirocin + Chlorhexidine | Education + Mupirocin + Bleach Baths
Number analyzed (Participants) | 64 | 62 | 64 | 54
Participants | 24 | 35 | 35 | 34

2. Secondary Outcome: Number of Participants With Recurrent Staphylococcus Aureus Skin or Soft Tissue Infection
Description: Recurrent Staphylococcus aureus Skin or Soft Tissue Infection is defined as incidence of skin abscess, impetigo, cellulitis, or spider bite in the 1 month following intervention. Infections reported by participant at follow-up visit.
Time Frame: 1, 4 and 6 month follow-ups
Population: Groups 1/4 have 1 more participant analyzed each than in participant flow module due to data collected by phone. They did not return to hospital for followup (colonization swabs were not obtained). Group 3 has 1 less participant analyzed than in participant flow module due to missing data point on followup survey. They were not able to be reached.
Measure: Number; unit: Participants
Arm/Group | 1: Hygiene Education | 2: Hygiene Education + Mupirocin | Education + Mupirocin + Chlorhexidine | 4: Education + Mupirocin + Bleach Baths
Number analyzed (Participants) | 65 | 62 | 63 | 55
Participants
  1 Month Follow-up | 17 | 14 | 7 | 12
  4 Month Follow-up | 26 | 20 | 19 | 18
  6 Month Follow-up | 28 | 27 | 23 | 21

3. Secondary Outcome: Number of Participants Eradicated of S. Aureus Carriage - 4 Months After Intervention
Description: as for outcome 1
Time Frame: 4 month follow-up
Measure: Number; unit: Participants
Arm/Group | 1: Hygiene Education | 2: Hygiene Education + Mupirocin | Education + Mupirocin + Chlorhexidine | 4: Education + Mupirocin + Bleach Baths
Number analyzed (Participants) | 64 | 57 | 57 | 51
Participants | 31 | 32 | 31 | 36

ADVERSE EVENTS:
Time Frame: Adverse events were collected by phone approximately 7-10 days following study enrollment. The intervention only lasted 5 days and thus all adverse events would have happened by this time.
Description: There are more participants with data on adverse events than data on the primary outcome measure because some participants completed the follow-up phone call at 7-10 days (where adverse events were assessed) but failed to complete the 1 month follow-up visit (where primary outcome measure was assessed).
Arm/Group | Hygiene Education | Hygiene Education + Mupirocin | Education + Mupirocin + Chlorhexidine | Education + Mupirocin + Bleach Baths
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/72 | 0/70 | 0/68
Other Adverse Events (participants affected / at risk) | 4/72 | 1/72 | 5/70 | 11/68
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Hygiene Education (N=72) | Hygiene Education + Mupirocin (N=72) | Education + Mupirocin + Chlorhexidine (N=70) | Education + Mupirocin + Bleach Baths (N=68)
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 1 | 5 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No